CLINICAL TRIAL: NCT02466789
Title: Investigating a Von Willebrand Factor (VWF) Functional Screening Assay for Assigning the Phenotypic Variants of Von Willebrand Disease (VWD)
Acronym: VWF-phV
Status: Completed | Type: Observational
Sponsor: Jonathan Roberts (Other)
Collaborators: Versiti Blood Health (Other)
Responsible Party: Sponsor-Investigator, Jonathan Roberts, Assistant Research Director, Bleeding and Clotting Disorders Institute Peoria, Illinois
Organization: Bleeding and Clotting Disorders Institute Peoria, Illinois (Other)
Other Study IDs: H14-25321
Record Dates: First submitted 2015-06-05; First posted 2015-06-09 (Estimated); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Von Willebrands Disease
Keywords: Bleeding Disorder, inherited; Von Willebrands Disease; Hematologic Test; VWF; VWD
MeSH Terms: conditions — von Willebrand Diseases; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sodium Citrated Plasma samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to improve the investigators ability to diagnose von Willebrand Disease (VWD), a common inherited bleeding disorder. This study will look at a new screening blood test used to determine if a person has VWD. This new screening blood test can determine a diagnosis more rapidly than current blood tests. Also this test could be available at local hospital labs rather than require samples to be sent to bigger more specialized labs.

DETAILED DESCRIPTION:
This investigation will be a prospective, multicenter trial to validate the clinical utility of a novel screening assay as a diagnostic screening assay for VWD variants: Type 1C, 2A, 2B, 2M and 2N. Once the subject is enrolled into the study, a minimum of 0.5ml of citrated plasma will be collected and analyzed at the Bleeding and Clotting Disorders Institute Laboratory in Peoria Illinois. Results will be collected: phenotype function profiles will be determined, statistically analyzed and compared to the qualitative data from Blood Center of Wisconsin. Data is expected to correlate as previously shown in prior studies and will confirm the utility of this assay.

ELIGIBILITY:
Inclusion Criteria:

* New subjects undergoing evaluation for the diagnosis of VWD determined to have a VWF:Ag or VWF: RCo < 50 IU/dl and or a VWF:RCo/VWF:Ag of <0.7. Also subjects will be included if Type 2 N VWD is clinically suspected

Exclusion Criteria:

* Those subjects whose lab results do not meet the inclusion criteria

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: New subjects undergoing evaluation for the diagnosis of VWD that are determined to have VWF:ag or VWF:RCo <50 IU/dl and or a VWF:RCo/VWF:ag ratio of <0.7. Also subjects will be included if Type 2N VWD is suspected
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2015-07; Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Validate the novel ELISA-based VWF functional screening assay as a diagnostic screening assay to assign VWD phenotypes 1C, 2A, 2B, 2M and 2N. | planned analysis at 2 years and 4 years with study duration estimated at 4 years

SECONDARY OUTCOMES:
Further development of the VWF functional screening assay through investigating the incorporation of VWF:CB6 (binding to collagen VI) | study duration 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Roberts, MD, Principal Investigator — Bleeding and Clotting Disorders Institute
Locations (1):
- Bleeding and Clotting Disorders Institute, Peoria, Illinois, United States

REFERENCES:
- [Background] Nichols WL, Hultin MB, James AH, Manco-Johnson MJ, Montgomery RR, Ortel TL, Rick ME, Sadler JE, Weinstein M, Yawn BP. von Willebrand disease (VWD): evidence-based diagnosis and management guidelines, the National Heart, Lung, and Blood Institute (NHLBI) Expert Panel report (USA). Haemophilia. 2008 Mar;14(2):171-232. doi: 10.1111/j.1365-2516.2007.01643.x. PMID 18315614
- [Background] Rodeghiero F, Castaman G, Dini E. Epidemiological investigation of the prevalence of von Willebrand's disease. Blood. 1987 Feb;69(2):454-9. PMID 3492222
- [Background] Werner EJ, Broxson EH, Tucker EL, Giroux DS, Shults J, Abshire TC. Prevalence of von Willebrand disease in children: a multiethnic study. J Pediatr. 1993 Dec;123(6):893-8. doi: 10.1016/s0022-3476(05)80384-1. PMID 8229521
- [Background] Werner EJ, Abshire TC, Giroux DS, Tucker EL, Broxson EH. Relative value of diagnostic studies for von Willebrand disease. J Pediatr. 1992 Jul;121(1):34-8. doi: 10.1016/s0022-3476(05)82537-5. PMID 1625090
- [Background] Castaman G, Eikenboom JC, Bertina RM, Rodeghiero F. Inconsistency of association between type 1 von Willebrand disease phenotype and genotype in families identified in an epidemiological investigation. Thromb Haemost. 1999 Sep;82(3):1065-70. PMID 10494765
- [Background] Rodeghiero F, Castaman G, Tosetto A. von Willebrand factor antigen is less sensitive than ristocetin cofactor for the diagnosis of type I von Willebrand disease--results based on an epidemiological investigation. Thromb Haemost. 1990 Nov 30;64(3):349-52. PMID 2096485
- [Background] Bazhan SV, Zhdanov VP, Koshil' OI. [Experience in organizing rehabilitative treatment for infectious patients]. Voen Med Zh. 1991 Jul;(7):35-6. No abstract available. Russian. PMID 1835556
- [Background] Castaman G, Tosetto A, Goodeve A, Federici AB, Lethagen S, Budde U, Batlle J, Meyer D, Mazurier C, Goudemand J, Eikenboom J, Schneppenheim R, Ingerslev J, Habart D, Hill F, Peake I, Rodeghiero F. The impact of bleeding history, von Willebrand factor and PFA-100((R)) on the diagnosis of type 1 von Willebrand disease: results from the European study MCMDM-1VWD. Br J Haematol. 2010 Nov;151(3):245-51. doi: 10.1111/j.1365-2141.2010.08333.x. Epub 2010 Aug 25. PMID 20738304
- [Background] Federici AB, Mannucci PM, Castaman G, Baronciani L, Bucciarelli P, Canciani MT, Pecci A, Lenting PJ, De Groot PG. Clinical and molecular predictors of thrombocytopenia and risk of bleeding in patients with von Willebrand disease type 2B: a cohort study of 67 patients. Blood. 2009 Jan 15;113(3):526-34. doi: 10.1182/blood-2008-04-152280. Epub 2008 Sep 19. PMID 18805962
- [Background] Federici AB, Canciani MT. Clinical and laboratory versus molecular markers for a correct classification of von Willebrand disease. Haematologica. 2009 May;94(5):610-5. doi: 10.3324/haematol.2009.005751. PMID 19407316